CLINICAL TRIAL: NCT02012335
Title: Ketamine Use in Electroconvulsive Therapy: Clinical, Cognitives and Neurotrophic Outcomes
Brief Title: Ketamine Use in Electroconvulsive Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Methodologicals and logistics issues.
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-0196
Record Dates: First submitted 2013-11-18; First posted 2013-12-16 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Electroconvulsive Therapy; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ECT + saline (Placebo Comparator): Brief pulse ECT with saline as placebo in each session
- ECT + Ketamine (Experimental): Brief pulse ECT with 0.05 mg/kg ketamine infusion in each session
  Interventions: Drug: ECT + Ketamine

INTERVENTIONS:
Drug: ECT + Ketamine — Brief pulse ECT with 0.05 mg/kg ketamine infusion in each session
  Arms: ECT + Ketamine

SUMMARY:
The purpose of this study is to determine whether combination of ketamine plus electroconvulsive therapy improves depressive symptoms decreasing cognitive side effects.

DETAILED DESCRIPTION:
This study will compare the clinical response to brief pulse ECT with infusion of ketamine 0.5 mg/kg versus brief pulse electroconvulsive therapy with infusion of placebo (saline) in major depression. We also will compare levels of cognitive impairment among these groups, compare levels of quality of life among these groups, compare levels of BDNF among these groups. We also will study if levels of 25-hydroxyvitamin D are associated with cognitive impairment in subjects undergoing ECT.

ELIGIBILITY:
Inclusion criteria

- Patients with unipolar and bipolar depression from The Psychiatric Unit of Hospital de Clinicas de Porto Alegre (diagnosis will be established by the Structured Clinical Interview for DSM-IV Axis I)

Exclusion criteria:

* Patients with dementia
* History of addiction / abuse of psychoactive drugs
* Other psychiatric diagnoses
* Refusal to follow the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale (HAM-D) 17 change | Baseline, week 1, week 2, week 3, week 4, and at the end of hospital stay, an expected average of 5 weeks

SECONDARY OUTCOMES:
Mini Mental Status Exam change | Baseline and at the end of hospital stay, an expected average of 5 weeks
Autobiographical Memory Test change | Baseline and at the end of hospital stay, an expected average of 5 weeks
Rey Auditory Verbal Learning Test change | Baseline and at the end of hospital stay, an expected average of 5 weeks
WAIS Digit Span change | Baseline and at the end of hospital stay, an expected average of 5 weeks
FAS verbal fluency change | Baseline and at the end of hospital stay, an expected average of 5 weeks
Stroop Test change | Baseline and at the end of hospital stay, an expected average of 5 weeks
Trial Making Test change | Baseline and at the end of hospital stay, an expected average of 5 weeks
WAIS Vocabulary | Baseline
Montgomery and Asberg Depression Rating Scale change | Baseline, week 1, week 2, week 3, week 4, and at the end of hospital stay, an expected average of 5 weeks
Brief Psychiatry Rating Scale change | Baseline, week 1, week 2, week 3, week 4, and at the end of hospital stay, an expected average of 5 weeks
Clinical Global Impression-Severity change | Baseline, week 1, week 2, week 3, week 4, and at the end of hospital stay, an expected average of 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Rio Grande do Sul / Hospital de Clínicas de Porto Alegre (HCPA), Porto Alegre, Rio Grande do Sul, Brazil